CLINICAL TRIAL: NCT05646121
Title: Post-market Clinical Follow-up Study to Evaluate the Performance and Safety of Suprasorb® A + Ag Wound Dressing and Rope in the Treatment of Wounds at Risk of Infection and Infected Wounds
Brief Title: Suprasorb® A + Ag in the Treatment of Wounds at Risk of Infection and Infected Wounds
Status: Completed | Type: Observational
Sponsor: Lohmann & Rauscher (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-02
Record Dates: First submitted 2022-09-19; First posted 2022-12-12 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pressure Ulcer; Arterial Ulcers; Venous Leg Ulcer; Diabetic Ulcers; Surgical Wound; Skin Graft
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wounds at risk of infection: Ideally 71 patients with wounds at risk of infection (W.A.R. Score ≥ 3) to be included.
  Interventions: Device: Suprasorb® A + Ag wound dressing and rope
- infected wounds: Ideally 28 patients with infected wounds (TILI Score ≥ 5) to be included.
  Interventions: Device: Suprasorb® A + Ag wound dressing and rope

INTERVENTIONS:
Device: Suprasorb® A + Ag wound dressing and rope — Suprasorb® A + Ag Antimicrobial Calcium Alginate Wound Dressings / Packing Rope are soft, conformable wound coverings with a high mannuronic acid content (mass per unit area ≥100 g/m2). The silver impregnated calcium alginate fibres react with wound exudate or blood to form a gel which creates a moist wound environment. The silver contained in the wound dressing has broad antimicrobial activity, including against MRSA and VRE. Antimicrobial action (>3 log steps) associated with the ionic silver from the silver alginate fibres (1.5%) is observed in vitro after just 24 h and this remains stable for up to seven days

SUMMARY:
The aim of this post market clinical follow up (PMCF) study is to confirm the performance of Suprasorb® A + Ag wound dressing and rope, to collect safety data regarding expected adverse events and to detect potential unexpected adverse events associated with use of Suprasorb® A + Ag wound dressing and rope within the certified indications and under the conditions of routine use.

DETAILED DESCRIPTION:
This clinical investigation will be conducted as 3 weeks, multicentre, open, single-arm cohort study on patients presenting wounds at risk of infection or infected wounds. All wounds of the included patients will be treated with Suprasorb® A +Ag Antimicrobial Calcium Alginate Wound Dressings (and Suprasorb® A + Ag Antimicrobial Calcium Packing Rope - if required by the depth of the wound).

At inclusion visit (V1, day 0), interim visit (V2, after 10 days ±3 days) and termination visit (V3 after 21 days ±3 days or earlier; as soon as the wound is epithelialized completely) patients will have clinical examination and wound area measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is legally capable
* Presence of a heavily exuding wound
* Presence of one of the following wounds:

  * pressure ulcers
  * arterial ulcers
  * venous lower leg ulcers
  * diabetic ulcers OR
  * postoperative wound
  * skin graft and donor sites
* Infected wound (TILI Score ≥ 5) or a wound with risk of infection (W.A.R. Score ≥ 3)
* Wound area between 4 and 100 cm2
* It must be possible to display the entire wound area on one photo from a distance of 25-30 cm
* Patient has signed a written Informed Consent

Exclusion Criteria:

* Treatment with Suprasorb® A + Ag Antimicrobial Calcium Algi-nate Wound Dressing and Rope or any silver containing dressing or topical drug during the last 3 weeks
* Known sensitivity to Suprasorb® A + Ag Antimicrobial Calcium Alginate Wound Dressing and Rope or any of their components
* Malignant wounds (tumor related wounds)
* Critical limb ischemia
* Infected wounds requiring systemic antibiotic therapy at baseline visit or infected wounds with surrounding skin requiring local an-tibiotics at baseline visit and/or during study conduct.
* Severe sensitive neuropathy (9-10 points on the Neuropathie-Symptom-Score (Diagnose und Therapie der sensomotorischen diabetischen Neuropathien. Diabetes und Stoffwechsel, 11, Suppl.2 (2002))
* Planned amputation within the next 1 months
* A planned surgical operation in the region of the study wound within the next 4 weeks following inclusion
* Patient is not compliant regarding treatment of the underlying disease (e.g. compression)
* Dry wound
* Pregnancy or breast feeding
* Reliable severe malnutrition
* Patient is analphabet
* Participation in any clinical trial within the last 1 month and during participation in this study
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main target population of this investigation are older people. Patients will be enrolled with wounds at risk of infection and infected wounds which are: heavily exuding, superficial or deep, for:
  * pressure ulcers
  * arterial ulcers
  * venous lower leg ulcers
  * diabetic ulcers
  * post-operative wounds
  * skin graft and donor sites.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Combined endpoint | 20 months
  Change of local wound infection after 21 days of treatment with Suprasorb® A+Ag in wounds at risk of infection and infected wounds, assessed by "Therapeutical Index for Local Infections (TILI)" score.
  The investigator will evaluate six indirect parameters of the local wound infection:
  * erythema to surrounding skin
  * heat
  * oedema, induration or swelling
  * spontaneous pain or pressure pain
  * stalled wound healing
  * increase and/or change in colour or smell of exudate
  Each present parameter will be assigned 1 point. All points will be summed up and the final score (min 0, max 6) will define the local infection status. In case the score is ≥ 5, wound is deemed to be locally infected.

SECONDARY OUTCOMES:
Rate of device-related adverse events (device safety) | 20 months
  Frequency and character severity of device deficiencies (DDs), adverse events (AEs), serious adverse events (SAEs), adverse device effects (ADEs), serious adverse device effects (SADEs) and incidents.
Change of wound bed condition, defined by the combination of the following parameters: | 20 months
  * Wound shift (reduction change of distribution of necrotic, fibrin and granulation tissue in % of the wound area), measured by W.H.A.T. (Wound Healing Analyzing Tool)
  * Wound shift (change of distribution of necrotic, fibrin and granulation tissue in % of the wound area), assessed visually by the investigators
  * Change in grade of exudation (from very high to none)
  * Change in type of exudate (from purulent to clear)
  * Change of peri-wound skin condition (presence or absence of erosion, maceration, dryness /scaling, edema, redness)
  * Wound size reduction over time measured by W.H.A.T. (Wound Healing Analyzing Tool)
  * Achieved healing rate, measured as a proportion of patients having complete wound epithelization after 20 months of treatment to the whole study population
Change in wound-related pain, with a separate assessment of: | 20 months
  * pain by dressing removal measured by NRS (numeric-rating scale from 0 to 10, where 0=no pain, 10=worst pain imaginable)
  * change in general wound related pain, measured by NRS (numeric-rating scale from 0 to 10, where 0=no pain, 10=worst pain imaginable)
Change in wound-related quality of life | 20 months
  Change in wound-related quality of life, measured by Wound QoL Questionnaire
User satisfaction | 20 months
  User satisfaction, assessed by the questionnaire
Mean frequency of dressing changes | 20 months
  Mean frequency of dressing changes
Mean time of treatment | 20 months
  Mean time of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Feldkamp, Dr., Study Director — Lohmann & Rauscher
Locations (8):
- Poland (8):
  - Private Practice, Bolesławiec
  - Private Practice, Krakow
  - Private Practice, Lodz
  - Private Practice, Ostróda
  - Private Practice, Oświęcim
  - Private Practice, Pabianice
  - Private Practice, Swidnica
  - Private Practice, Wroclaw

IPD SHARING:
Plan to Share IPD: No